CLINICAL TRIAL: NCT05161650
Title: Modulation of Circulating Levels of the Ketone Body 3-hydroxybutyrate in Patients With Chronic Heart Failure: Cardiovascular Effects
Brief Title: Hemodynamic Effects of Chronic Ketosis.
Acronym: KETO-CHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristoffer Berg-Hansen, Principal Investigator, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KETO-CHF
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone monoester (3-OHB) (Experimental)
  Interventions: Dietary Supplement: Ketone monoester (3-OHB)
- Isocaloric placebo (Experimental)
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Ketone monoester (3-OHB) — Commercially available ketone supplement
  Arms: Ketone monoester (3-OHB)
Dietary Supplement: Placebo drink — Isocaloric placebo
  Arms: Isocaloric placebo

SUMMARY:
Heart Failure (HF) is a major public health issue because the disease affects 1-2% of the Western population and the lifetime risk of HF is 20%. Despite major improvements in the management and care of patients with HF, the 1-year mortality in patients with HF is 13% and >50% of HF patients are admitted during a 2.5 year period. Furthermore, patients with HF have markedly decreased physical capacity and quality of life. Thus, there is a need for new treatment modalities in this group of patients.

We have shown, using positron emission tomography, that ketone body infusion reduces myocardial glucose uptake and increases myocardial blood flow in healthy subjects. Data from another study conducted by our group show a 40% increase in cardiac output during infusion of 3-OHB in patients with HF and reduced left ventricular ejection fraction (HFrEF).

Presently there are no data on the clinical cardiovascular effects of long-term oral ketone-supplementation in patients with chronic HF.

In this study we aim to investigate the effect of 14 days modulation of circulating ketone body levels on cardiac function and exercise capacity in patients with HFrEF.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure with NYHA II-III
* Left ventricular ejection fraction ≤40%
* Negative urine-HCG for women with childbearing potential

Exclusion Criteria:

* Known diabetes or HbA1c ≥48 mmol/mol
* Significant cardiac valve disease
* Severe stable angina pectoris
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Resting cardiac output (L/min) | 14 days of dietary supplement
  Measured with right heart catheterization

SECONDARY OUTCOMES:
Resting pulmonary capillary wedge pressure (PCWP) | 14 days of dietary supplement
  Measured with right heart catheterization
Peak exercise pulmonary capillary wedge pressure (PCWP) | 14 days of dietary supplement
  Measured with right heart catheterization
Peak exercise cardiac output (L/min) | 14 days of dietary supplement
  Measured with right heart catheterization
Exercise capacity (METs) | 14 days of dietary supplement
  Cardiopulmonary exercise test

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Berg-Hansen K, Gopalasingam N, Christensen KH, Ladefoged B, Andersen MJ, Poulsen SH, Borlaug BA, Nielsen R, Moller N, Wiggers H. Cardiovascular Effects of Oral Ketone Ester Treatment in Patients With Heart Failure With Reduced Ejection Fraction: A Randomized, Controlled, Double-Blind Trial. Circulation. 2024 May 7;149(19):1474-1489. doi: 10.1161/CIRCULATIONAHA.123.067971. Epub 2024 Mar 27. PMID 38533643